CLINICAL TRIAL: NCT03370848
Title: A Prospective Randomized, Open-Label, Crossover Study on the Effects of Psyllium on Niacin Tolerability
Brief Title: Effects of Psyllium on Niacin Tolerability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 039
Record Dates: First submitted 2016-12-20; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Flushing; Hyperlipidemias; Dyslipidemias
Keywords: Niacin; Psyllium; Dietary fiber
MeSH Terms: conditions — Flushing; Hyperlipidemias; Dyslipidemias | interventions — Psyllium; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psyllium plus Aspirin and Niacin ER (Experimental): Niacin ER 500mg tablet - take 1 niacin ER 500mg tablet at least two hours before bedtime for two weeks, then increase niacin ER to two 500mg tablets (1,000 mg total) for two weeks, then increase to three niacin ER 500mg tablets (1,500 mg total) for two weeks.
  Aspirin 325mg tablet - take 1 aspirin 325 mg tablet 30 minutes prior to niacin ER
  Psyllium 1.7gm wafers - take 2 wafers (3.4 grams total) along with aspirin 30 minutes prior to niacin ER
  Interventions: Dietary Supplement: Psyllium; Drug: Aspirin
- Aspirin and Niacin ER (Active Comparator): Niacin ER 500mg tablet - take 1 niacin ER 500mg tablet at least two hours before bedtime for two weeks, then increase niacin ER to two 500mg tablets (1,000 mg total) for two weeks, then increase to three niacin ER 500mg tablets (1,500 mg total) for two weeks.
  Aspirin 325mg tablet - take 1 aspirin 325 mg tablet 30 minutes prior to niacin ER
  Interventions: Drug: Aspirin

INTERVENTIONS:
Dietary Supplement: Psyllium — Aspirin 325 mg tablet and two 1.7gm psyllium wafers (3.4gm total) 30 minutes prior to niacin ER
  Other Names: Metamucil; Cilium; Fiberall
  Arms: Psyllium plus Aspirin and Niacin ER
Drug: Aspirin — Aspirin 325 mg tablet 30 minutes prior to niacin ER
  Other Names: Bayer; Ecotrin

SUMMARY:
The purpose of this study is to determine whether psyllium is effective in reducing flushing due to niacin and also to measure the effect of niacin on cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are starting ER niacin for clinical indication by a healthcare provider
* No prior use of psyllium for the past 2 months
* No prior use of niacin for the past 3 months
* Ability to give informed consent
* Must be reachable by telephone

Exclusion Criteria:

* Known contraindications to ER niacin, aspirin or psyllium (including: presence of nausea, vomiting, abdominal pain, intestinal obstruction, or fecal impaction; known hypersensitivity to ER niacin, aspirin or psyllium; severe hepatic dysfunction, transaminitis; history of gastrointestinal bleed attributable to aspirin induced gastritis)
* Patient who are unable to perform assessment of flushing using the standardized scales or questionnaires
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Global Flushing Severity Score | up to 6 weeks

SECONDARY OUTCOMES:
HDL | Baseline, & end of week 6
LDL | Baseline, & end of week 6

CONTACTS AND LOCATIONS:
Overall Officials: Freny V Mody, MD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (1):
- VA West Los Angeles Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No